CLINICAL TRIAL: NCT04479579
Title: Towards Improved Adherence With Extended Venous Thromboembolism Prophylaxis After Abdominal or Pelvic Major Cancer Surgery
Brief Title: Improved Adherence With Extended Venous Thromboembolism Prophylaxis After Major Cancer Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sam Schulman, Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10768
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Neoplasms Malignant; Surgery; Venous Thromboembolism; Prophylaxis; Adherence, Medication
Keywords: apixaban; abdominal; pelvic
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apixaban (Experimental): apixaban for extended prophylaxis against VTE after discharge
  Interventions: Drug: Apixaban 2.5 milligram

INTERVENTIONS:
Drug: Apixaban 2.5 milligram — apixaban 2.5 milligram twice daily from discharge until postoperative day 29 +/- 1 day
  Other Names: medication adherence assessment

SUMMARY:
This is a prospective, twin-center, cohort study in patients discharged from the hospital after major abdominal or pelvic cancer surgery for cancer. This study is designed to evaluate the adherence to extended deep vein thrombosis prophylaxis (DVT) with the direct oral anticoagulant apixaban on the background of historical data from the investigator's center on low-molecular-weight heparin (LMWH) substandard adherence in the same setting.

DETAILED DESCRIPTION:
All guidelines have embraced the concept of extended DVT prophylaxis after major abdominal or pelvic surgery for cancer, but the recommendation is consistently to use LMWH, which is more complicated than orally available prophylaxis, more expensive and has poor adherence.

The patients will be identified in the pre-operative admission or in post-operative orders as potentially eligible for extended prophylaxis. On the day of discharge a research assistant or a research nurse will approach the patient, provide information about the study and obtain written consent if the patient fulfills the eligibility criteria.

Each patient will be asked to take apixaban until postop day 29±1 and will be followed until postop day 90±3. The total duration of the study from first patient in to last patient out is expected to take 12 months.

At 1 week after discharge there is a telephone contact to ask about any side effects from apixaban or bleeding events or signs of thromboembolism and to answer any questions from the patient.

At postoperative Day +28-30 there is a telephone contact to ask about side effects, bleeding, signs of venous thromboembolism (VTE), until what date the patient has taken apixaban and estimate of missed doses using a standardized script. If the patient is still taking it, instruction will be given to discontinue. Self-reported modified Morisky Medication Adherence scale with 6 statements will be used At 90 days ±3 days there is the last telephone contact to ask about bleeding events or signs of VTE. The study is complete for the patient. At the time of Visit 4 the pharmacy that the patient uses will be contacted to provide dispensing record for apixaban, in order to verify that the patient filled the prescription.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years of age, discharged after hepato-biliary, colorectal or gynecology-oncology abdominal/pelvic surgery (laparoscopic or open) for cancer and considered at increased risk for VTE (e.g. previous history of VTE, residual cancer, slow mobilization, obesity, comorbidities).
* Written informed consent obtained.

Exclusion Criteria:

* Patient unable to take tablets, even if crushed.
* Active bleeding.
* Venous thromboembolism diagnosed during the hospitalization.
* Severe hepatic impairment (Child Pugh class C).
* Severe renal failure on dialysis or with calculated creatinine clearance <15 mL/min.
* Platelet count <50·109/L.
* Concomitant treatment with azole-antimycotics, e.g., ketoconazole, itraconazole, voriconazole, or posaconazole, and HIV protease inhibitors, e.g., ritonavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male, female, other
Enrollment: 53 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Filled prescription | 1 week
  Percent of included patients that have filled their prescription for apixaban
At least 80% adherence | 30 days
  Percent of patients with filled prescription that have at least 80% adherence

SECONDARY OUTCOMES:
Rate of Venous thromboembolism post prophylaxis | 2 months
  The event rate of venous thromboembolism during the 2 months after planned prophylaxis

OTHER OUTCOMES:
Rate of Venous thromboembolism during prophylaxis | 30 days
  Symptomatic, objectively verified deep vein thrombosis of pulmonary embolism during 1st month
Rate of Major bleeding during prophylaxis | 30 days
  Major bleeding during 1st month
Rate of Clinically relevant non-major bleeding during prophylaxis | 30 days
  Clinically relevant non-major bleeding during 1st month
Rate of Death during prophylaxis | 30 days
  Death during 1st month

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, MD, PhD, Principal Investigator — Dr.
Locations (2):
- Canada (2):
  - Thrombosis Service, HHS-General Hospital, Hamilton, Ontario
  - HHS-Juravinski Hospital, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serrano PE, Parpia S, Valencia M, Simunovic M, Bhandari M, Levine M. Incidence of delayed venous thromboembolic events in patients undergoing abdominal and pelvic surgery for cancer: a systematic review and meta-analysis. ANZ J Surg. 2019 Oct;89(10):1217-1223. doi: 10.1111/ans.15290. Epub 2019 Jun 18. PMID 31210407
- [Background] Serrano PE, Parpia S, Linkins LA, Elit L, Simunovic M, Ruo L, Bhandari M, Levine M. Venous Thromboembolic Events Following Major Pelvic and Abdominal Surgeries for Cancer: A Prospective Cohort Study. Ann Surg Oncol. 2018 Oct;25(11):3214-3221. doi: 10.1245/s10434-018-6671-7. Epub 2018 Jul 26. PMID 30051364
- [Result] Schulman S, Carlson V, Serrano PE, Sne N, Kahnamoui K, Mithoowani S, Ikesaka R, Gross PL. Adherence to apixaban for extended thromboprophylaxis after major abdominal or pelvic surgery for cancer: A prospective cohort study. J Surg Oncol. 2022 Aug;126(2):386-393. doi: 10.1002/jso.26876. Epub 2022 Apr 1. PMID 35362102
- See also: Publication of the study — https://pubmed.ncbi.nlm.nih.gov/35362102/